CLINICAL TRIAL: NCT01353989
Title: Hepatitis A Vaccination in the Elderly
Status: Completed | Type: Observational
Sponsor: Rijnstate Hospital (Other)
Responsible Party: dr EH Gisolf, Rijnstate Hospital, Arnhem, the Netherlands
Other Study IDs: Hepatitis A vaccination
Record Dates: First submitted 2010-06-21; First posted 2011-05-16 (Estimated); Last update posted 2016-06-28 (Estimated); Status verified 2016-06

CONDITIONS: Hepatitis A
Keywords: hepatitis A; vaccination; elderly; protection to hepatitis A after vaccination
MeSH Terms: conditions — Hepatitis A

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — 5 times 7 ml of blood will be collected
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- >60 years
- < 40 years

SUMMARY:
A lot of elderly people travel to hepatitis A endemic areas. The prevalence of hepatitis A IgG positivity is declining in the Netherlands, also in the elderly. Studies show that people above 40 years of age have a slower immune response to hepatitis A vaccination. However, a lot of travelers seek pre-travel advice only shortly before their journey. More information about the time to adequate antibody response after hepatitis A vaccination is required to provide good protection during travelling. Alternative protection with immunoglobulins are available.

Study design: Observational, longitudinal pilot study Study population: 20 adults over 60 years of age with a negative hepatitis A IgG, (with a estimated 50% positivity for hepatitis A IgG in this age Group, 40 patients in this age group) 20 adults 18-40 years of age as controls.

Intervention (if applicable): When hepatitis A vaccination is indicated and informed consent is obtained, hepatitis A IgG wil be measured at day 0, 7, 14, 21 en 28.

Main study parameters/endpoints: Time to protective hepatitis A IgG. Nature and extent of the burden and risks associated with participation, benefit and group relatedness: hepatitis A vaccination will be given also outside this study. In the study 5 venous punctures of 7 ml of blood.

ELIGIBILITY:
Exclusion Criteria:

* previous hep A vaccination
* known hepatitis A serology status
* immunodeficiency

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 80 >60 years, hepatitis A vaccination indicated 40 < 40 years, hepatitis A vaccination indicated
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2010-07; Primary Completion 2015-07 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
How fast do patients> 60 year reach protective anti-HAV levels after vaccination? | 0, 1,2,3,4 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Rijnstate Hospital, Arnhem, Netherlands